CLINICAL TRIAL: NCT03372616
Title: coMparison Between invAsive and Non-invasive assessmenT on Blood Pressure and Cardiac Function in HealthY Participants: the MATCHY Study
Brief Title: coMparison Between invAsive and Non-invasive assessmenT on Blood Pressure and Cardiac Function in HealthY Participants
Acronym: MATCHY
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Chief director of department of cardiology, Shanghai 10th People's Hospital
Other Study IDs: MATCHY2017YZ
Record Dates: First submitted 2017-10-29; First posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Healthy Volunteer
Keywords: aortic blood pressure; diastolic dysfuntion; echocardiography; left ventricular ejection fraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: Aortic blood pressure, LV filling pressrue, and LV volume will be measured in all participants. Meanwhile, echocardiography and non-invasive aortic blood presure measurement will be performed. Three devices will be used in non-invasive aortic blood presure measurement, including Sphygmocor (AtCor Medical, Australia), PulsePen (DiaTecne SRL, Italy), and Mobil-O-Graph (IEM, Germany). In conclusion, all participants will receive invasive and non-invasive left ventricular diastolic function assessment, together with invasive and non-invasive aortic blood pressure assessment.
  Interventions: Diagnostic Test: Invasive left ventricular diastolic function assessment; Diagnostic Test: Invasive aortic blood pressure measurement; Diagnostic Test: Non-Invasive left ventricular diastolic function assessment; Diagnostic Test: Non-Invasive aortic blood pressure measurement

INTERVENTIONS:
Diagnostic Test: Invasive left ventricular diastolic function assessment — Left ventricular (LV) polyethylene catheter was inserted into left ventricular to directly measure LV filling pressure.
Diagnostic Test: Invasive aortic blood pressure measurement — Aortic blood pressure will be measured with polyethylene catheter in aortic root.
Diagnostic Test: Non-Invasive left ventricular diastolic function assessment — Echocardiography will be performed in all participants to assess left ventricular diastolic function non-invasively.
Diagnostic Test: Non-Invasive aortic blood pressure measurement — Three devices (Sphygmocor [AtCor Medical, Australia], PulsePen [DiaTecne SRL, Italy], and Mobil-O-Graph [IEM, Germany] ) will be used to assess aortic blood pressure non-invasively when participants are undergoing invasive aortic blood pressure measurement.

SUMMARY:
This is a cross-sectional cohort study which aims to compare the invasive and non-invasive assessments on aortic blood pressure and cardiac funtion in subjects without history of cardio-vascular disease. Left ventricular (LV) filling pressure, LV volume, and aortic blood pressure will be measured invasively. Non-invasive assessment includes echocardiography,aortic, and carotid blood pressure measurement.

ELIGIBILITY:
Inclusion Criteria:

* Over or equal to 18 years old;
* Agree to participate the study and sign informed written consent;
* Any change of drugs which effect the hemodynamics during 1 month prior to enrollment;
* Proposed to perform coronary angiography and left left ventriculography in hospital;

Exclusion Criteria:

* Non-sinus rhythm or frequent extra systoles;
* Identified coronary artery disease via coronary angiography;
* Diagnosed pulmonary vascular or parenchymal disease;
* Hypertrophic cardiomyopathy, restrictive cardiomyopathy, or constrictive pericarditis;
* Stenosis or insufficiency of valves (moderate and above);
* Heart transplant;
* Congenital heart disease;
* Inadequate imaging or doppler parameter quality in echocardiography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with proposed coronary angiography and left left ventriculography but without diagnosed cardiovascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Left ventricular filling pressure assessment with left heart catheterization | 1 day
  All participants will receive invasive left ventricular filling pressure assessment with left heart catheterization.
Left ventricular diastolic function assessment with echocardiography using ASE recommendations | 1 day
  All participants will receive non-invasive left ventricular diastolic function assessment with echocardiography. The ASE-recommended (American Society of Echocardiography) creteria would be used to define left ventricular diastolic dysfunction.
Left ventricular diastolic function assessment with echocardiography using EACVI recommendations | 1 day
  All participants will receive non-invasive left ventricular diastolic function assessment with echocardiography. The EACVI-recommended (European Association of Cardiovascular Imaging) creteria would be used to define left ventricular diastolic dysfunction.

SECONDARY OUTCOMES:
Aortic blood presure obtained with Sphygmocor device | 1 day
  Sphygmocor device (AtCor Medical, Australia) will be used in non-invasive aortic blood presure measurement with standard protocols shown in its user manual.
Aortic blood presure obtained with PulsePen device | 1 day
  PulsePen device (DiaTecne SRL, Italy) will be used in non-invasive aortic blood presure measurement with standard protocols shown in its user manual.
Aortic blood presure obtained with Mobil-O-Graph device | 1 day
  Mobil-O-Graph (IEM, Germany) device will be used in non-invasive aortic blood presure measurement with standard protocols shown in its user manual.
Aortic blood presure obtained with catheterization | 1 day
  Catheterization will be used in invasive aortic blood presure measurement. The cather will be placed in the aortic root while measuring the blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Yawei Xu, M.D., Ph.D., Study Chair — Shanghai 10th People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagueh SF, Smiseth OA, Appleton CP, Byrd BF 3rd, Dokainish H, Edvardsen T, Flachskampf FA, Gillebert TC, Klein AL, Lancellotti P, Marino P, Oh JK, Popescu BA, Waggoner AD. Recommendations for the Evaluation of Left Ventricular Diastolic Function by Echocardiography: An Update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2016 Apr;29(4):277-314. doi: 10.1016/j.echo.2016.01.011. No abstract available. PMID 27037982
- [Background] Handoko ML, Paulus WJ. Polishing the diastolic dysfunction measurement stick. Eur J Echocardiogr. 2008 Sep;9(5):575-7. doi: 10.1093/ejechocard/jen181. Epub 2008 Jun 11. No abstract available. PMID 18579489
- [Background] McEniery CM, Cockcroft JR, Roman MJ, Franklin SS, Wilkinson IB. Central blood pressure: current evidence and clinical importance. Eur Heart J. 2014 Jul;35(26):1719-25. doi: 10.1093/eurheartj/eht565. Epub 2014 Jan 23. PMID 24459197